CLINICAL TRIAL: NCT01165944
Title: Effectiveness of Pramlintide on Control of Post-Transplant Diabetes Mellitus
Brief Title: Effectiveness Study of Pramlintide to Treat Post-Transplant Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1343
Record Dates: First submitted 2010-06-09; First posted 2010-07-20 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus
Keywords: Post transplant diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard diabetes therapy (No Intervention): Standard diabetes therapy with either oral agents or insulin injections
- Oral diabetic agents and pramlintide (Active Comparator)
  Interventions: Drug: Pramlintide
- Insulin injection with pramlintide (Active Comparator)
  Interventions: Drug: Pramlintide

INTERVENTIONS:
Drug: Pramlintide — Pramlintide administered pre-meal starting at 60 mcg and titrating up to 120 mcg within 4-6 weeks
  Arms: Insulin injection with pramlintide; Oral diabetic agents and pramlintide

SUMMARY:
Post-transplant diabetes mellitus (PTDM) develops in up to 30% of patients undergoing solid organ transplantation. This disease is difficult to treat as the levels of glycemia fluctuate in response to variations in doses of steroid and other immunosuppressive agents. At the same time, poorly controlled hyperglycemia affects negatively graft function and survival as well as on the ability of the immunocompromised host to fight infections. The investigators hypothesize that the addition of Pramlintide (Symlin) to the management of patients with PTDM would help patients with post-transplant diabetes attain better control at the critical time of titration of immunosuppressive regimens. The primary objective of this proposal is to improve glycemic control of diabetes with Pramlintide in patients with post-transplant diabetes at 3 and 6 months of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Post-transplant diabetes (PTMD)
* Aged 20-70
* Diagnosis of diabetes within the last 6-18 months
* Stable medications
* Stable weight for 3 months
* Serum creatinine < 1.5 mg/dL

Exclusion Criteria:

* Pre-transplant diabetes
* Major postoperative complications following transplant
* Pregnancy
* Significant GI discomfort with nausea or vomiting
* Inability to learn continuous glucose monitoring
* Development of diabetes more than 4 years after transplant
* omen of child-bearing potential who use birth control pills and have fasting triglycerides of > 400 mg/dL

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
HgA1c | 6 months
  Primary outcomes utilized in this study will be endpoints of HbA1C

SECONDARY OUTCOMES:
Continuous glucose monitoring | 6 months
  Secondary outcomes will include mean blood glucose levels assessed by continuous glucose monitoring (CGM) at 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris Draznin, M.D., Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States